CLINICAL TRIAL: NCT00338975
Title: Cognitive Behavioral Skills Training for Schizophrenia
Brief Title: Cognitive Behavioral Social Skills Training for Improving Social Functioning in People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eric L. Granholm, Professor of Psychiatry, UCSD, San Diego Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH071410 (NIH); R01MH071410 (NIH); DSIR 83-ATAP (Other: NIMH/DSIR)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia
Keywords: Psychotic Disorders; Schizoaffective Disorder; Cognitive Behavioral Therapy; Social Skills Training
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Organizational Objectives

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cognitive Behavioral Social Skills Training (CBSST)
  Interventions: Behavioral: Cognitive Behavioral Social Skills Training (CBSST); Behavioral: Social Skills Training; Behavioral: Goal Setting
- 2 (Active Comparator): Goal-Focused Supportive Contact (GFSC)
  Interventions: Behavioral: Goal-focused supportive contact (GFSC); Behavioral: Goal Setting

INTERVENTIONS:
Behavioral: Cognitive Behavioral Social Skills Training (CBSST) — There are 36 weekly group sessions, each session is 2 hours in length, with a half-hour break after the first hour. The intervention integrates CBT and SST techniques and neurocognitive compensatory aids. All participants are asked to identify a goal. The SST components are based, in part, on a pre-packaged SST intervention available from Psychiatric Rehabilitation Consultants. The CBT components are based on techniques developed for CBT in general and techniques developed specifically for patients with schizophrenia. Cognitive therapy is combined with role-play practice of communication skills and problem-solving training.
  Other Names: CBT; SST
  Arms: 1
Behavioral: Goal-focused supportive contact (GFSC) — There are 36 weekly group sessions, each 2 hours in length, with a half-hour break after the first hour. GFSC has a number of specific goals and interventions, including providing a safe environment where the patient can discuss her/his feelings and concerns; to validate these feelings and concerns; and to provide support and guidance to the client so that she/he can make progress to solving problems or alleviating concerns and worries. Psychotic symptoms and cognition are not directly targeted. Therapists utilize "non-specific" therapeutic techniques, including providing unconditional positive regard, reflective listening, encouraging, paraphrasing, and summarizing. Therapists do not develop a formulation or teach skills.
  Arms: 2
Behavioral: Social Skills Training — The SST components are based, in part, on a pre-packaged SST intervention available from Psychiatric Rehabilitation Consultants. Participants engage in role plays and problem solving.
  Other Names: SST
  Arms: 1
Behavioral: Goal Setting — All participants are asked to identify a personally meaningful goal as soon as possible in therapy. Over the 36 weeks, participants in CBSST learn skills related to goal attainment, while participants in GFSC do not receive skills aimed at goal attainment, but are encouraged to discuss their goals .

SUMMARY:
This study evaluated the effectiveness of Cognitive Behavioral Social Skills Training versus goal-focused supportive contact in improving social functioning in people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic, severe, and disabling brain disorder. People with schizophrenia sometimes hear voices others don't hear, believe that others are broadcasting their thoughts to the world, or become convinced that others are plotting to harm them. These symptoms make it difficult for people with schizophrenia to interact normally and establish healthy social relationships with others. Cognitive Behavioral Social Skills Training (CBSST) is a group behavioral therapy intervention that focuses on improving cognitive and metacognitive impairments and social skills deficits that interfere with normal functioning in people with schizophrenia. Goal-focused supportive contact (GFSC) is a group therapy intervention that focuses on helping people with schizophrenia to verbalize their problems or worries and to seek advice from fellow group members. This study evaluated the effectiveness of CBSST versus GFSC in improving social functioning in people with schizophrenia. The study will assessed changes in cognition, psychotic symptoms, and use of psychiatric healthcare services.

Participants in this open label study were randomly assigned to one of the following treatment groups: treatment as usual (TAU) plus CBSST or TAU plus GFSC. Both interventions consist of 2-hour therapy sessions weekly for 36 weeks. Groups receiving each intervention do not exceed ten people. CBSST integrates cognitive therapy, social skills training, and neurocognitive compensatory aids. Cognitive therapy helps participants challenge unhelpful thoughts and build communication and problem-solving skills. Participants receive workbooks that describe the skills and contain homework assignments. GFSC focuses on empowering participants to share problems, worries, or concerns with others who face similar issues. Participants share advice with each other, but therapists do not teach skills. Outcomes were be assessed at Months 4.5, 9, 15, and 21 for all participants.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder at any stage of illness

Exclusion Criteria:

* Level of care required at baseline interferes with outpatient group therapy participation (e.g., partial or inpatient hospitalization for psychiatric illness, substance use, or physical illness)
* No case manager or care coordinator
* Medically or psychiatrically unstable for outpatient therapy
* Exposure to social skills training (SST), cognitive behavioral therapy (CBT), or dialectical behavioral therapy (DBT) within 5 years prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2005-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Social Functioning | Measured at baseline and Months 9 and 21
  Independent Living Skills Survey (ILSS), PSR Toolkit, Maryland Assessment of Social Competence (MASC)

SECONDARY OUTCOMES:
Neuropsychological functioning | Measured at baseline and Months 9 and 21
  Delis-Kaplan Executive Function System (D-KEFS; 20 Questions, Card Sort, Word Context), Trails A & B, Letter Number Sequencing, Wechsler Memory Scale (WMS) Spatial Span, Hopkins Verbal Learning Test (HVLT), Brief Visuospatial Memory Test (BVMT)
Cognitive insight | Measured at baseline and Months 4.5, 9, 15, and 21
  Birchwood Insight Scale, Beck Cognitive Insight Scale
Psychotic symptoms | Measured at baseline and Months 4.5, 9, 15, and 21
  Positive and Negative Syndrome Scale (PANSS), Psychotic Symptoms Rating Scales (PSY-RATS), Paranoia Scale, Beliefs About Voices Questionnaire (BAVQ-R)

CONTACTS AND LOCATIONS:
Overall Officials: Eric L. Granholm, PhD, Principal Investigator — VA San Diego Healthcare System/University of California San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Background] Granholm E, McQuaid JR, McClure FS, Auslander LA, Perivoliotis D, Pedrelli P, Patterson T, Jeste DV. A randomized, controlled trial of cognitive behavioral social skills training for middle-aged and older outpatients with chronic schizophrenia. Am J Psychiatry. 2005 Mar;162(3):520-9. doi: 10.1176/appi.ajp.162.3.520. PMID 15741469
- [Background] Granholm E, McQuaid JR, McClure FS, Pedrelli P, Jeste DV. A randomized controlled pilot study of cognitive behavioral social skills training for older patients with schizophrenia. Schizophr Res. 2002 Jan 1;53(1-2):167-9. doi: 10.1016/s0920-9964(00)00186-9. No abstract available. PMID 11728848
- [Background] McQuaid JR, Granholm E, McClure FS, Roepke S, Pedrelli P, Patterson TL, Jeste DV. Development of an integrated cognitive-behavioral and social skills training intervention for older patients with schizophrenia. J Psychother Pract Res. 2000 Summer;9(3):149-56. PMID 10896740
- [Background] Brenner HD, Hodel B, Genner R, Roder V, Corrigan PW. Biological and cognitive vulnerability factors in schizophrenia: implications for treatment. Br J Psychiatry Suppl. 1992 Oct;(18):154-63. No abstract available. PMID 1389037
- [Background] Granholm E, McQuaid JR, McClure FS, Link PC, Perivoliotis D, Gottlieb JD, Patterson TL, Jeste DV. Randomized controlled trial of cognitive behavioral social skills training for older people with schizophrenia: 12-month follow-up. J Clin Psychiatry. 2007 May;68(5):730-7. doi: 10.4088/jcp.v68n0510. PMID 17503982
- [Derived] Granholm E, Holden J, Link PC, McQuaid JR. Randomized clinical trial of cognitive behavioral social skills training for schizophrenia: improvement in functioning and experiential negative symptoms. J Consult Clin Psychol. 2014 Dec;82(6):1173-85. doi: 10.1037/a0037098. Epub 2014 Jun 9. PMID 24911420